CLINICAL TRIAL: NCT06551675
Title: A Randomized, Double-blind, Very Low Dose Parallel-controlled, Prospective, Multi-center Trial Evaluating the Improvement of Nutritional Status and Frailty With Silkworm Pupa Tablets After Radical Resection of Gastrointestinal Malignancies
Brief Title: Effect of Silkworm Pupa Tablets in Gastrointestinal Malignancies at Nutritional Risk Following Radical Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xiaosun Liu, MD (Other)
Responsible Party: Sponsor-Investigator, Xiaosun Liu, MD, Deputy director of gastrointestinal surgery department, First Affiliated Hospital of Zhejiang University
Organization: First Affiliated Hospital of Zhejiang University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IIT20240064C
Record Dates: First submitted 2024-08-06; First posted 2024-08-13 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Nutritional Deficiency; Gastrointestinal Cancer; Frailty Syndrome
Keywords: silkworm pupa tablets; gastrointestinal malignancies; nutritional risk; frailty
MeSH Terms: conditions — Malnutrition; Gastrointestinal Neoplasms; Frailty | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Silkworm pupa tablets group (Experimental): Wanshililongbao silkworm pupa tablets.
  Interventions: Dietary Supplement: Silkworm pupa tablets
- Control group (Sham Comparator): Contains 0.5% of the active ingredient of the study product, indistinguishable in appearance.
  Interventions: Dietary Supplement: Control product

INTERVENTIONS:
Dietary Supplement: Silkworm pupa tablets — Participants will begin taking the silkworm pupa tablets immediately upon enrollment, 1200mg/tablet, two tablets a time, twice a day (BID), with a treatment duration of three months.
  Arms: Silkworm pupa tablets group
Dietary Supplement: Control product — The sham comparator contains 0.5% of the active ingredient of the study product, indistinguishable in appearance. Participants will begin taking the control immediately upon enrollment, 1200mg/tablet, two tablets a time, twice a day (BID), with a treatment duration of three months.
  Arms: Control group

SUMMARY:
This is a randomized, double-blind, very low dose parallel-controlled, prospective, multi-center trial evaluating the improvement of nutritional status and frailty with silkworm pupa tablets after radical resection of gastrointestinal malignancies for 3 months intervention. The primary endpoints are body weight and frailty prevalence, The secondary endpoints are body mass index (BMI), skeletal muscle index (SMI) at the third lumbar vertebra (L3-SMI), sarcopenia prevalence and quality of life.

DETAILED DESCRIPTION:
Previous study has indicated that silkworms pupae extracts may increase muscle mass and strength, here we conduct a randomized, double-blind, very low dose parallel-controlled, prospective, multi-center trial.

1. Study population: malignant gastrointestinal tumors, including gastric cancer, colorectal cancer, esophageal cancer, and pancreatic cancer, and has undergone radical surgical resection. If necessary, perioperative systemic treatment has been completed by the time of screening, and has a nutritional risk score of ≥3 (based on the NRS 2002 nutritional risk screening tool).
2. Sample size: totally 120 cases, including 60 cases in the experimental group and 60 cases in the control group.
3. Research content: In this study, participants will begin taking the trial product or control immediately upon enrollment, with a treatment duration of 3 months.Experimental Group: Wanshililongbao silkworm pupa tablets. Control Group: contains 0.5% of the active ingredient of the trial product, indistinguishable in appearance.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily participate in the clinical study, fully understand the study and sign the informed consent form (ICF); willing and able to follow and complete all trial procedures.
* Gender unrestricted, age at the time of signing ICF: ≥18 years, ≤80 years.
* Diagnosed with a malignant gastrointestinal tumor, including gastric cancer, colorectal cancer, esophageal cancer, and pancreatic cancer, and has undergone radical surgical resection. If necessary, perioperative systemic treatment has been completed by the time of screening.
* At the time of screening, a nutritional risk score of ≥3 (based on the NRS 2002 nutritional risk screening tool) .
* In good general condition, with an ECOG performance status score of ≤2.
* Agree to provide peripheral blood, stool, and urine samples for biomarker analysis during the study period.

Exclusion Criteria:

* At the time of screening, presence of tumor recurrence or metastasis.
* At the time of screening, presence of another active malignancy requiring concurrent treatment.
* Expected survival of ≤3 months.
* Unable to take oral nutrition, requiring enteral feeding tubes, or having malabsorption syndrome or any condition affecting gastrointestinal absorption; e.g., chronic diarrhea (watery stools; defecation frequency ≥5 times a day).
* Patients who are planning a pregnancy, are pregnant, or are breastfeeding.
* Allergic to any known components of the trial materials.
* Presence of serious primary diseases of the heart, brain, lungs, liver, kidneys, endocrine, hematological, neurological, or other systems, or other acute or chronic diseases that could significantly affect treatment and prognosis.
* Presence of other severe physical or mental illnesses or laboratory abnormalities that may increase the risk associated with participation in the study, or patients deemed unsuitable for participation by the researchers.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2024-08-14 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Body weight | 3 months
  Measured at baseline and 1 month, 2 months, 3 months after enrollment
Frailty prevalence | 3 months
  The incidence of frailty, using Fried frailty phenotype to assess physical frailty, measured at baseline and 1 month, 2 months, 3 months after enrollment

SECONDARY OUTCOMES:
Body mass index (BMI) | 3 months
  Calculated as weight (kg)/height (m2), measured at baseline and 1 month, 2 months, 3 months after enrollment
L3-SMI | 3 months
  Derived as the ratio of skeletal muscle area (SMA) to height [SMA (cm2)/height (m2)], at the third lumbar vertebra, measured at baseline and after 3 months
Sarcopenia prevalence | 3 months
  The incidence of sarcopenia, using the diagnostic criteria for sarcopenia published by the Asian Sarcopenia Working Group (AWGS) in 2019 or L3-SMI criteria, measured at baseline and 1 month, 2 months, 3 months after enrollment
Quality of life | 3 months
  Using the questionnaire of EORTC QLQ-C30 measured at baseline and 1 month, 2 months, 3 months after enrollment
Quality of life | 3 months
  Using the questionnaire of EORTC QLQ-STO22, measured at baseline and 1 month, 2 months, 3 months after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Xiaosun Liu, Principal Investigator — First Affiliated Hospital of Zhejiang University
Locations (4):
- China (4):
  - Affiliated Hangzhou First People's Hospital, School of Medicine, Westlake University, Hangzhou, Zhejiang
  - The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - The Second Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - Hangzhou Institute of Medicine Chinese Academy of Sciences, Hangzhou

IPD SHARING:
Plan to Share IPD: No